CLINICAL TRIAL: NCT03435484
Title: Using Rapid Cycle Randomized Controlled Trials to Increase Completion Rates of the Patient-Reported Health Assessment Questionnaire During Outpatient Visits at NYU Langone Orthopedic Center
Brief Title: Using RCT to Increase Completion Rates of the Health Assessment Questionnaire.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RCT PHA Optimization
Record Dates: First submitted 2018-01-23; First posted 2018-02-19 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Patient-reported Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Participants in this group will receive one version (out of two) of instructions for completing the Health Assessment Questionnaire.
  Interventions: Other: Arm A
- Arm B (Active Comparator): Participants in this group will receive another version (out of two) of instructions for completing the Health Assessment Questionnaire.
  Interventions: Other: Arm B

INTERVENTIONS:
Other: Arm A — Intervention includes various iterations of instructions for completing the Health Assessment Questionnaire. Participants in this group will receive one version (out of two) of instructions for completing the Health Assessment Questionnaire.
  Arms: Arm A
Other: Arm B — Intervention includes various iterations of instructions for completing the Health Assessment Questionnaire. Participants in this group will receive another version (out of two) of instructions for completing the Health Assessment Questionnaire.
  Arms: Arm B

SUMMARY:
The proposed study aims to examine several iterations of instructions/reminders that patients receive for completing the Health Assessment Questionnaire (self-reported health outcomes) for their outpatient visit at NYU Langone Orthopedic Center. The goal is to increase the completion rates of patient-reported health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are eligible to receive the Health Assessment Questionnaire in preparation for and during their outpatient visit to the NYU Langone Orthopedic Center.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27263 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire Completion Rate (number of times patients complete or partially complete the questionnaire). | Duration of the study, up to 6 months.
  Completion rate data is routinely collected by the medical center.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States